CLINICAL TRIAL: NCT05402488
Title: Exploring the Recovery Function of Sleep in Neurodegeneration - an Observational Cross-Sectional Study
Brief Title: Exploring the Recovery Function of Sleep in Neurodegeneration
Acronym: RFSN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RFSN
Record Dates: First submitted 2021-12-21; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Neurodegenerative Diseases
Keywords: Parkinson's Disease; Huntington's Disease; MCI; Neurodegenerative Diseases; Sleep; Auditory Stimulation
MeSH Terms: conditions — Neurodegenerative Diseases; Parkinson Disease; Huntington Disease | interventions — Acoustic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: During data collection, participants will be blinded to the condition, i.e. sham or verum stimulation. All experimenters will be blind for processing and analysis of outcome measures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum stimulation (Experimental): Verum condition: Auditory stimulation during sleep
  Interventions: Behavioral: Auditory stimulation
- Sham stimulation (Sham Comparator): Sham condition: Playing no tones during sleep but still recording brain activity (muted tones)
  Interventions: Behavioral: Auditory stimulation

INTERVENTIONS:
Behavioral: Auditory stimulation — Auditory stimulation during sleep

SUMMARY:
The overall objective of this study is to identify the best approach for assessing the recovery function of sleep in neurodegenerative diseases associated with abnormal protein aggregation with regard to the conception of future intervention studies. To this end, the investigators will follow an exploratory approach in a preferably broad data set collected in patients with neurodegenerative diseases associated with abnormal protein aggregation and in healthy humans.

DETAILED DESCRIPTION:
First, the investigators want to assess the relationship between sleep parameters (e.g. sleep intensity) and behavioral/cognitive performance and subjective measures (e.g. sleep quality, mood, and sleepiness) in patients with neurodegenerative disorders associated with abnormal protein aggregation. Healthy subjects will be assessed for procedure validation and reference purposes. Second, the investigators want to probe whether associations can be influenced by modulation of sleep parameters by means of auditory stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Good general health or confirmed diagnosis of neurodegenerative disease associated with abnormal protein aggregation along international criteria
* Age above 18 years
* In ambulant setting: ability to apply the ambulant EEG device for the duration of the study, either alone or with help of co-habitant if MoCA < 20

Exclusion Criteria:

* Failure to give informed consent
* Inability to follow the procedures of the study, e.g. due to language problems or cognitive deficits
* Known or suspected non-compliance, drug- or medication abuse
* Inability to hear the tones to be applied during sleep in auditory stimulation experiments
* Skin disorders/problems/allergies in face/ear area that could worsen with electrode application
* Regular intake of drugs that may alter the relationship between sleep and outcome variables under investigation (opioids, benzodiazepines and z-drugs (nonbenzodiazepines)).
* Clinically significant concomitant disease states
* Too high (disease) burden for patients
* Additional non-medical exclusion criteria may be defined for certain cognitive tasks (e.g. no glasses during experiments involving eye tracking)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Electrophysiological markers of brain activity during sleep as measured with EEG | measured during 4 nights
  e.g. slow wave activity (SWA)
Performance change in behavioral/cognitive tasks | measured before and after 4 nights
  e.g. reaction time
Change in outcomes of subjective measures | measured before and after 4 nights
  e.g. sleepiness (scale from 1 to 10)

SECONDARY OUTCOMES:
Outcomes of other physiological measures during sleep | measured during 4 nights
  e.g. muscle activity (EMG)
Outcomes of other physiological measures during behavioral tasks | measured before and after 4 nights
  e.g. pupil dilation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Neurology department, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No